CLINICAL TRIAL: NCT07258550
Title: Effects of the Otago Exercise Programme on Senior Physical Fitness, Balance, and Quality of Life Among Older Adults in Sarawak: A Randomised Controlled Trial
Brief Title: Otago Exercise Programme and Physical Function in Older Adults in Sarawak
Acronym: OEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Malaysia Sarawak (Other)
Responsible Party: Principal Investigator, Anselm Ting Su, Professor, Faculty of Medicine & Health Sciences, Universiti Malaysia Sarawak (UNIMAS), University Malaysia Sarawak
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UNIMAS-OEP-2024; SELF-FUNDED-DRPH-2024 (Other Grant/Funding Number: Dr Saravanan Muruthamuthu (self-funded DrPH))
Record Dates: First submitted 2025-11-17; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Accidental Falls; Balance Assessment; Physical Fitness
Keywords: Otago Exercise Programme; Balance; Physical fitness; Quality of life; Older adults; Sarawak; Fall prevention; Community-dwelling elderly

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into two parallel groups: an intervention group receiving the Otago Exercise Programme (OEP) and a control group continuing their usual daily activities without structured exercise. Both groups were followed for 12 weeks with assessments at baseline, 6 weeks, and 12 weeks.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Triple-blind randomized controlled trial. Participants, investigators, and outcome assessors were blinded to group allocation. Randomization codes were generated and maintained by an independent coordinator until completion of all data collection and analyses to prevent bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Otago Exercise Programme (OEP) (Experimental): Participants in the intervention group will receive the Otago Exercise Programme (OEP), a structured, multicomponent home- and group-based exercise programme focusing on lower-limb strength, balance, and functional mobility. Each supervised session lasts about 60 minutes and includes warm-up, strengthening, balance, and cool-down exercises. Sessions are conducted three times weekly for 12 weeks under supervision by trained facilitators, with participants encouraged to continue selected exercises at home.
  Interventions: Behavioral: Otago Exercise Programme (OEP)
- No Intervention: Usual Daily Activity (Control) (No Intervention): Participants in the control group will continue their usual daily activities and will not participate in any structured exercise programme. They will receive general health education leaflets on physical activity and fall prevention at baseline, without additional supervised training.

INTERVENTIONS:
Behavioral: Otago Exercise Programme (OEP) — The Otago Exercise Programme (OEP) is a behavioural, multicomponent exercise protocol focusing on lower-limb strength, balance, and functional mobility. It includes warm-up, strengthening, balance, and cool-down components performed three times weekly for 12 weeks under trained supervision. The programme aims to improve balance, enhance lower-limb strength, and reduce fall risk among community-dwelling older adults.
  Arms: Experimental: Otago Exercise Programme (OEP)

SUMMARY:
This randomized controlled trial aims to evaluate the effects of the Otago Exercise Programme (OEP) on physical fitness, balance, and quality of life among older adults in Sarawak, Malaysia. The intervention involves a structured home-based and group-supervised exercise programme focused on lower-limb strength and balance training. A total of 120 community-dwelling older adults aged 60 years and above were recruited from Bau District, Sarawak, and randomized into intervention (OEP) and control groups. The intervention group participated in the OEP for 12 weeks, while the control group maintained their usual activities.

Assessments were conducted at baseline, 6 weeks, and 12 weeks using the Senior Fitness Test (SFT), Berg Balance Scale (BBS), and WHOQOL-BREF to evaluate changes in physical fitness, balance, and quality of life. The study aims to provide evidence on the effectiveness of OEP as a feasible, community-based fall-prevention and functional fitness programme for older adults in Malaysia. Findings will contribute to national healthy ageing policy and rehabilitation strategies under the WHO Decade of Healthy Ageing (2021-2030) framework.

DETAILED DESCRIPTION:
This study used a two-arm, parallel-group randomized controlled trial design to evaluate the effectiveness of the Otago Exercise Programme (OEP) in improving physical fitness, balance, and functional mobility among community-dwelling older adults in the Bau District of Sarawak, Malaysia.

Participants were screened for eligibility and safety using clinical history, medical clearance forms, and physical readiness questions. Randomization was conducted using computer-generated permuted blocks, with allocation sequences prepared and concealed by an independent coordinator not involved in assessment or intervention delivery.

The intervention protocol followed the standardized OEP training manual and included lower-limb strengthening, balance exercises, functional mobility tasks, and progressive walking prescriptions. Participants performed three weekly home-based sessions supported by weekly group-supervised sessions led by trained facilitators. Exercise progression was individualized according to participant capability and safety guidelines.

Outcome assessments were conducted at baseline, week 6, and week 12 by assessors who were blinded to group allocation. Standardized measurement procedures were used following the Senior Fitness Test (SFT) manual and the Berg Balance Scale (BBS) assessment protocol. Adverse events and training adherence were monitored throughout the intervention period.

The study operated under ethical approval from the Medical Research Ethics Committee, Universiti Malaysia Sarawak (Ref: FME/24/115). This project was conducted as part of a Doctor of Public Health (DrPH) research requirement. Findings are expected to contribute evidence for community-based fall-prevention strategies and healthy ageing programmes in Malaysia.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling older adults aged 60 to 100 years residing in Bau District, Sarawak.
* Able to ambulate independently, with or without an assistive device.
* Physically and cognitively able to participate in exercise sessions.
* Willing to provide written informed consent and commit to the 12-week programme and all scheduled assessments.
* Medically cleared for moderate-intensity exercise by a healthcare provider.

Exclusion Criteria:

* Severe visual, auditory, neurological, or musculoskeletal impairment that limits safe participation in exercise.
* Unstable medical conditions (e.g., uncontrolled hypertension, recent cardiac event, severe respiratory illness).
* Cognitive impairment or diagnosed dementia preventing informed participation.
* Currently participating in any other structured exercise or physiotherapy programme.
* Any contraindication to moderate-intensity physical activity as determined by screening or medical history.

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Balance performance measured using the Berg Balance Scale (BBS) | Baseline, 6 weeks, and 12 weeks after intervention start
  Balance ability will be assessed using the Berg Balance Scale (BBS), a 14-item objective measure designed to evaluate balance in older adults. Each item is scored on a 5-point scale (0-4), with a total possible score of 56. Higher scores indicate better balance and lower fall risk.

SECONDARY OUTCOMES:
30-Second Chair Stand Test Performance | Baseline, 6 weeks, and 12 weeks after intervention start
  The 30-second chair stand test will assess lower-body strength. Participants will be instructed to stand up fully and sit down as many times as possible within 30 seconds. Higher scores represent greater lower-body strength.
Arm Curl Test Performance | Baseline, 6 weeks, and 12 weeks after intervention start
  Upper-body strength will be assessed using the Arm Curl Test. Participants will perform as many arm curls as possible in 30 seconds using a standardized dumbbell (5 lbs for women and 8 lbs for men). A higher number of repetitions indicates greater upper-body strength.
2-Minute Step Test Performance | Baseline, 6 weeks, and 12 weeks after intervention start
  Aerobic endurance will be assessed using the 2-minute step test. Participants will march in place for 2 minutes, lifting the knees to a height midway between the patella and iliac crest. The number of steps meeting the required height will be counted. Higher numbers indicate greater aerobic endurance.
Chair Sit-and-Reach Test Performance | Baseline, 6 weeks, and 12 weeks after intervention start
  Flexibility will be assessed using the chair sit-and-reach test. Participants will sit on the edge of a chair with one leg extended and reach toward the toes. The distance reached (positive score for reaching past the toes, negative score if short of toes) will be recorded. Higher values indicate better lower-body flexibility.
Back Scratch Test Performance | Baseline, 6 weeks, and 12 weeks after intervention start
  Upper-body flexibility will be assessed using the back scratch test. Participants will place one hand over the shoulder and the other behind the back, attempting to touch or overlap the middle fingers. The distance between the fingertips (positive score for overlap, negative for gap) will be recorded. Higher values indicate better upper-body flexibility.
8-Foot Up-and-Go Test Performance | Baseline, 6 weeks, and 12 weeks after intervention start
  Agility and dynamic balance will be assessed using the 8-foot up-and-go test. Participants will rise from a seated position, walk 8 feet, turn around, and return to sit down as quickly as possible. The total time taken (in seconds) will be recorded. Shorter times indicate better agility and dynamic balance.

OTHER OUTCOMES:
Quality of life measured using the WHOQOL-BREF questionnaire | Baseline, 6 weeks, and 12 weeks after intervention start
  Quality of life will be assessed using the World Health Organization Quality of Life-BREF (WHOQOL-BREF) questionnaire, which consists of 26 items covering four domains: physical health, psychological well-being, social relationships, and environment. Higher domain scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Dewan Tasik Biru, Bau, Sarawak, Malaysia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared because the dataset contains identifiable information related to community-dwelling older adults in Sarawak. Data access is restricted under the Universiti Malaysia Sarawak (UNIMAS) Medical Ethics Committee approval. Only aggregated or anonymized results will be available upon reasonable request to the corresponding author.